CLINICAL TRIAL: NCT01510756
Title: A Phase II Translational Study of Sorafenib for the Treatment of Chronic Lymphocytic Leukemia Patients
Brief Title: Sorafenib for the Treatment of Chronic Lymphocytic Leukemia (CLL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Thomas Kipps (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Thomas Kipps, Professor of Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110574
Record Dates: First submitted 2012-01-11; First posted 2012-01-16 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Experimental): Sorafenib 400mg orally twice daily will be administered for three cycles (1 cycle = 28 days).
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 400mg orally twice daily will be administered for three cycles (1 cycle = 28 days). Subjects without significant toxicity or progressive disease may elect to continue treatment for a total of twelve cycles.
  Other Names: Nexavar

SUMMARY:
This is a Phase 2 trial to evaluate the activity of sorafenib in relapsed or refractory CLL patients with an iwCLL-WG indication to receive therapy.

Sorafenib is an orally active multikinase inhibitor, which targets the RAF/MEK/ERK signaling pathway as well as several receptor tyrosine kinases. It is FDA approved for the treatment of hepatocellular carcinoma and renal cell carcinoma. Preclinical studies in the investigators laboratory demonstrated that sorafenib is cytotoxic to CLL cells.

The primary objective of the study is to determine the overall response rate of Sorafenib in previously treated CLL patients. All patients will receive sorafenib at 400 mg twice daily continuously for three months and then assessed for response. Responding patients may elect to continue on treatment for an additional 9 months.

DETAILED DESCRIPTION:
The UCSD Moores Cancer is conducting a Phase 2 clinical trial to evaluate the activity of sorafenib in relapsed or refractory CLL patients.

Sorafenib (BAY 43-9006) is an oral multi-kinase inhibitor with effects on tumor proliferation and tumor angiogenesis. It was initially selected based on inhibition of the serine/threonine kinases Raf-1 and wild-type B-Raf, which are pivotal components of the Ras/Raf/MEK/ERK signaling pathway. CLL cells derive survival support from their microenvironment, in part by activation of this pathway. Preclinical studies performed in our lab demonstrated that sorafenib was cytotoxic to CLL cells, including those from patients with more aggressive disease and from patients with chemotherapy (fludarabine) resistant disease.

The purpose of this study is to evaluate for evidence of anti-leukemic activity / clinical activity of sorafenib by assessing decrease in absolute lymphocyte count (ALC)/leukemia cell counts, lymphadenopathy, splenomegaly, and leukemia infiltration of bone marrow and to assess the impact of sorafenib on the CLL B cells through corollary studies. Patients will continue treatment for up to 3 monthly cycles unless toxicity or progressive disease. Patients with noted stable disease (or better) in the absence of significant toxicity will be allowed to receive another 1-9 cycles of single agent sorafenib. All patients will be assessed for response following 3 cycles of treatment and/or following all therapy per iwCLL-WG 2008 guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed or refractory CLL.
* Experiencing progressive disease with an iwCLL-WG indication to receive therapy.
* Age ≥ 18 years.
* ECOG performance status ≤ 2 at study entry.
* Adequate organ and marrow function as defined below:
* platelets ≥ 50 x 109/L
* serum creatinine ≤ 1.5 mg/dL
* total bilirubin ≤ 1.5 mg/dL
* AST(SGOT)/ALT(SPGT) ≤ 2 X institutional upper limit of normal or if known liver involvement <5X institutional upper limit of normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* No investigational agents within 28 days prior to entering the study.
* No concurrent use of other anti-cancer agents or treatments.
* No congestive heart failure > class II NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (beginning within the last 3 months) or myocardial infarction within the past 6 months.
* No known brain metastases (progressive neurologic dysfunction may confound the evaluation of neurologic and other adverse events).
* No cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* No uncontrolled hypertension defined as systolic blood pressure > 140 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* No known active Hepatitis or HIV.
* No history of allergic reactions attributed to compounds sorafenib or its excipients.
* No uncontrolled intercurrent illness such as ongoing or active infection (fungal, bacterial, and/or viral), CTCAE grade 2 or greater.
* No thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* No serious non-healing wound, ulcer, or bone fracture.
* No major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* No condition that may impair the patient's ability to swallow whole pills.
* Patient must not have any malabsorption problem.
* Patients receiving St. John's Wort or rifampin (rifampicin) are ineligible.
* Patients with uncontrolled Autoimmune Hemolytic Anemia (AIHA) or autoimmune thrombocytopenia (ITP) are ineligible.
* Patients must not be experiencing psychiatric illness/social situations that would limit compliance with study requirements.
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Subjects with any previously untreated or concurrent cancer that is distinct in primary site or histology from CLL except cervical cancer in-situ, treated basal cell carcinoma, squamous cell carcinoma of the skin, or superficial bladder tumor (Ta and Tis). Subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before study entry are allowed. All cancer treatments must be completed at least 3 years prior to study entry (ie, signature date of the informed consent form).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-12; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Kipps, M.D., Ph.D., Principal Investigator — UCSD Medical Center
Locations (1):
- UCSD Medical Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sorafenib
Started | 4
Completed | 0
Not Completed | 4
Not completed — Death | 1
Not completed — Lack of Efficacy | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Determination of absolute lymphocyte count (ALC), lymphadenopathy, splenomegaly, and/or marrow leukemia as measured by 4-color flow minimal residual disease (MRD) panel after 3 cycles of study treatment. (Decrease in absolute lymphocyte count by 50%, decrease in lymphadenopathy (sum of lymph node product) by 50%, decrease in splenomegaly by 50%, or decrease in leukemia infiltration of the bone marrow by 50%.)
Time Frame: 3 months
Population: Zero participants analyzed due to termination of study
Arm/Group | Sorafenib
Number analyzed (Participants) | 0

2. Secondary Outcome: To Determine the iwCLL-WG Defined Overall Response Rate (ORR) - Complete Response (CR) and Partial Responses (PR) to 3 Cycles of Sorafenib Therapy and Following the Completion of All Therapy.
Description: A response assessment must be performed 2 months following completion of therapy to document responses, including a bone marrow if in clinical response (CR) and a computed tomography (or magnetic resonance imaging scan [MRI]) if initial imaging was abnormal or physical examination inconclusive.
Time Frame: Two months following completion of treatment with sorafenib according to iwCLL guidelines.
Population: zero participants analyzed due to termination of study
Arm/Group | Sorafenib
Number analyzed (Participants) | 0

3. Secondary Outcome: Safety and Tolerability
Description: Frequency, severity and relatedness of adverse events
Time Frame: 3 months
Population: zero participants analyzed due to termination of study
Arm/Group | Sorafenib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Sorafenib
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=4)
Brain abscess (aspergillus) (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=4)
Abdominal pain (Gastrointestinal disorders) | 1
alopecia (Skin and subcutaneous tissue disorders) | 1
Amylase elevation (Metabolism and nutrition disorders) | 1
anorexia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 2
Hand foot syndrome (Skin and subcutaneous tissue disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
hyperbillirubinema (Hepatobiliary disorders) | 1
Lipase elevation (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Polyuria (Renal and urinary disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
neutropenia (Blood and lymphatic system disorders) | 1
thrombocytopenia (Blood and lymphatic system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes